CLINICAL TRIAL: NCT05134831
Title: Functional Medical Rhinoplasty: Objective Evaluation of the Efficacy of Hyaluronic Acid Injections in the Septo-triangular Angle in the Treatment of Internal Nasal Valves
Brief Title: Medical Rhinoplasty: Evaluation of the Efficacy of Hyaluronic Acid in the Treatment of Internal Nasal Valves.
Acronym: Rhinomedifon
Status: Withdrawn | Type: Observational
Why Stopped: issue reglementary
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0929
Record Dates: First submitted 2021-10-27; First posted 2021-11-26 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Nasal Obstruction
MeSH Terms: conditions — Nasal Obstruction | interventions — Rhinomanometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Rhinomanometry — At Day 0, before the hyaluronic acid injection, the patient's nasal breathing is assessed by 4-phase rhinomanometry (bilaterally: right nostril AND left nostril).
  At Month 1, the patient's nasal breathing is re-assessed by 4-phase rhinomanometry, in the same conditions as Day 0.

SUMMARY:
Nasal obstruction is a possible complication of rhinoplasty surgery. Several causes can explain it: deviation of the nasal septum, appearance of mucosal flanges inside the nasal cavity, but also collapse of the internal valve by its fragility. All surgeons performing rhinoplasty or rhinoseptoplasty are unfortunately confronted with this. Thus, when a rhinoplasty patient complains of postoperative nasal obstruction, the surgeon routinely performs several explorations:

* Inspection of the nasal cavity with a nasofibroscope
* Study of the nasal respiratory flows with a rhinomanometer The results of these 2 explorations allow to determine the cause of the obstruction and if it is explained or not by a collapse of the internal valve.

When internal valve collapse is the cause of postoperative nasal obstruction, few alternatives exist to treat this problem. Revision surgery under general anesthesia is usually necessary, with placement of a cartilage graft (= spreader graft) in the septo-triangular angle to reopen and support it. An alternative treatment is the injection of hyaluronic acid into the septo-triangular angle instead of the cartilage graft placed in the operating room. This option has several advantages: it is performed during the consultation, no general anesthesia is required, the procedure is quick, the cost is much lower, the patient's nasal breathing improves immediately, and the post-procedure follow-up is simple. The aim of our study is therefore to objectively analyze the modification of nasal biomechanics after injection of hyaluronic acid in the septo-triangular angle in patients with internal nasal valve (post (septo)-rhinoplasty). This objective evaluation will be performed with a rhinomanometer, before and after injection. This is a simple, non-invasive measuring device that allows the measurement of the main physical variables governing the biomechanics of the fluids inside the nasal cavity, such as pressure, flow and therefore nasal resistance. The objective proof of such an efficiency will allow a better management of the patients, to universalize the practices, to decrease the cost of the treatment and eventually to bring arguments to the health authorities for the reimbursement of such procedures.

ELIGIBILITY:
Inclusion Criteria:

* Major patients of all ages:
* Previous rhinoplasty or rhinoseptoplasty surgery
* Carrier of a nasal obstruction by collapsed internal valve
* Requiring an injection of hyaluronic acid in the septo-triangular angle
* Nasal obstruction by internal valve collapse is defined by (all elements must be present):
* Patient complaining of nasal obstruction (uni or bilateral)
* Collapse of the internal valve during normal nasal inspiratory effort on physical examination
* Improvement of the collapse and therefore of the nasal obstruction at the Bachmann maneuver during the physical examination
* Rhinomanometric internal valve criteria: area under the curve value on the flow/pressure diagram at the inspiratory phase ABOVE the diagnostic threshold (>18 622)
* Patients who did not object to their participation in the study

Exclusion Criteria:

1. Patients unable to complete questionnaires and visual scales
2. Patients with another cause of associated nasal obstruction:

   * Persistent septal deviation
   * Mucosal synechiae
   * Septal perforation
   * Turbinate hypertrophy
   * Inspiratory collapse of the external valve
   * Allergic rhinitis
   * Vasomotor rhinitis
   * Nasosinus polyposis
   * Nasal cavity or cavum tumors

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults Patients presenting a nasal obstruction post (septo)rhinoplasty, caused by an internal valve syndrome, which must benefit from an injection of hyaluronic acid will be included (in the absence of criteria of non-inclusion and after collection of the non-opposition of the patient).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Area under the curve of the "inspiratory open loop" on the flow-pressure diagram | change between Day 0 before injection and Month 1 after injection
  Value of the area of the "inspiratory open loop" (on the flow/pressure diagram produced by the rhinomanometer, in the inspiratory phase), and position of this value in relation to the diagnostic threshold of internal valve syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Alain-Ali MOJALLAL, MD, Principal Investigator — Service de chirurgie plastique, esthétique et reconstructrice